CLINICAL TRIAL: NCT02586818
Title: Clinical Performance of the Investigational InRhythm PT/INR System in a Professional Use Setting
Brief Title: Clinical Performance of Investigational InRhythm PT/INR System in a Professional Use Setting
Status: Withdrawn | Type: Observational
Why Stopped: Product was discontinued.
Sponsor: Accriva Diagnostics (Industry)
Collaborators: University of Rochester (Other)
Responsible Party: Sponsor
Other Study IDs: INR_CSP_015_0002_RA
Record Dates: First submitted 2015-10-22; First posted 2015-10-26 (Estimated); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Blood Dyscrasia
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Biospecimen Retention: Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is designed to evaluate and verify the clinical accuracy of the InRhythm PT/INR system; a point-of-care, whole blood PT/INR measurement with a reference plasma based PT/INR using a laboratory reference instrument and reagent (Sysmex/lnnovin) calibrated to the WHO rTF09 reference standard.

ELIGIBILITY:
Inclusion Criteria - All

* The subjects must be > 18 years of age.
* The subjects must be willing and competent to sign an informed consent.
* The subjects must be able to attend the clinic for one visit to donate one FS blood sample and one venous blood draw of approximately 10 cc.

Exclusion Criteria - All

* The subject is unable to donate fingerstick and venous blood samples.
* The subject has a history of clinically significant bleeding associated with incising the finger and/or the venipuncture.
* The subject is enrolled in any other study that involves an investigational drug and/or device.

Additional Inclusion Criteria - Therapeutic Group

* The subject must require oral VKA anticoagulant therapy.
* The patient must have been anticoagulated for at least three months prior to enrollment.

Additional Exclusion Criteria - Normal Group

- Subjects receiving any form of anticoagulation drugs such as Aspirin or Clopidogrel.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population to be studied consists of subjects who require oral anticoagulant therapy with VKA in accordance with the approved label indications for VKA administration. Normal healthy individuals will also be enrolled to collect data to support the low end of the lnRhythm system detection range.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Primary Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of INR measurements | 5 weeks